CLINICAL TRIAL: NCT04794543
Title: Effects of E-Cigarettes on the Lung Metabolome in People Living With HIV
Brief Title: Effects of Using E-Cigarettes on Lungs in People With HIV (HBS Ancillary)
Acronym: HBS Ancillary
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Director Clinical Nutrition and Metabolism Lab, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-028; U54GM104940 (NIH)
Record Dates: First submitted 2021-03-04; First posted 2021-03-12 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hiv; Lung Injury
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — breath samples, blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- e-cigarettes and/or e-liquid vaping smokers: actively use e-cigarettes or vape
- cigarette smokers: actively smoke combustible tobacco and/or marijuana (cannabis)
- Non-smokers: no use of e-cigarettes or vape or active smoking in the past 5 years (and less than a total of 10 pack-years lifetime use)

SUMMARY:
This is an ancillary study, thus participants will be recruited from participants in the HBS Study. This project acutely assesses the role of the e-cigarettes and vaping on lung health. The proposed work will inform the design of future studies to better understand vaping's health consequences and to test novel interventions to mitigate vaping's contribution to acute and/or chronic lung injury.

ELIGIBILITY:
This project is an ancillary study to the HBS Study. Inclusion Criteria for that IRB approved study are:

* documented HIV-infection
* in care at an HIV specialty clinic
* age ≥ 18 years.

Exclusion criteria for the HBS Study are:

* a pacemaker or other implanted electronic device
* pregnant women, prisoners, cognitively-impaired subjects.

For this ancillary, the experimental group must actively use at least one of the following: e-cigarettes, e-liquid vapes, burning leaf tobacco cigarettes, or inhaled burning leaf marijuana (cannabis). The control group will have no use of e-cigarettes or vape or active smoking in the past year.

Participants must be willing to archive data and biological samples for future use.

Exclusion from the ancillary are:

* overt respiratory or oral cavity disease
* acute illness in the past 4 weeks
* active cancer
* active weight loss program
* any other medical, psychiatric or behavioral factors that, in the judgment of the PI may interfere with study participation or ability to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV (PLWH) in the study site areas who are enrolled in the HBS study (main trial).
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Changes in respiratory tract metabolite profiles in PLWH | Baseline only (at Visit 1)
  Metabolomic analyses of exhaled breath condensate and gas.

CONTACTS AND LOCATIONS:
Overall Officials: John Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Lsuhsc-No, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No